CLINICAL TRIAL: NCT03255343
Title: Treatment of Non-responding to Conventional Therapy Inoperable Liver Cancers by in Situ Introduction of ImDendrim "[188Re]Rhenium Complex Coupled to an Imidazolic Ligand and Associated With a Dendrimer"
Brief Title: Treatment of Non-responding to Conventional Therapy Inoperable Liver Cancers by in Situ Introduction of ImDendrim
Acronym: ImDendrim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: French Association for the Advancement Medical Research (Other)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFPREMED
Record Dates: First submitted 2017-08-08; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Efficacy and Safety

STUDY DESIGN:
Intervention Model Description: 10 patients with liver tumor non operable, with resistance to other classical chemotherapy, injected a single dose of IMDENDRIM 10 mCi per 1 cm²
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMDENDRIM (Experimental)
  Interventions: Device: IMDENDRIM

INTERVENTIONS:
Device: IMDENDRIM — In situ and intra tumoral injection of non removal nanodevice IMDENDRIM

SUMMARY:
Objective (s) : To Evaluate the efficacy and safety of Treatment of non-responding to conventional therapy inoperable liver cancers by in situ introduction of ImDendrim.

Trial Design:

An, open-labeled and unicenter study in women or men with primary hepatocellular cancer or metastatic liver without standard therapeutic options for treatment including chemotherapy or surgery.

DETAILED DESCRIPTION:
Objective (s) : To Evaluate the efficacy and safety of Treatment of non-responding to conventional therapy inoperable liver cancers by in situ introduction of ImDendrim "[188Re] rhenium complex coupled to a imidazolic ligand and associated with a dendrimer".

Trial Design:

1. Type of the clinical Trial:

   An, open-labeled and unicenter study in women or men with primary hepatocellular cancer or metastatic liver without standard therapeutic options for treatment including chemotherapy or surgery.
2. Duration and method The trial will be comprised of 12 weeks of continued observation following in situ injection of ImDendrim into a subject suffering non-responding to conventional therapy inoperable liver cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have given written informed consent.
2. Female or male aged 18 years and over.
3. Confirmed histological diagnosis of primary hepatocellular cancer or metastatic liver without standard therapeutic options for treatment including chemotherapy or surgery. Not more than 5 measurable lesions at least 20 mm in the longest diameter by spiral Computed Tomography (CT) scan. Patients with hepatic tumor extended without discontinuity to regional structures are accepted (including vascular axis, lymphatic nodes and others organs namely pancreas, billiary vesicle and peritonea).
4. Life expectancy of 12 weeks or longer.
5. Patient with no contraindication to local anaesthesia.
6. Karnofsky index ≥ 70%
7. Negative pregnancy test for women of childbearing potential. -
8. Women should be under effective contraceptive method during at least trial period

Exclusion Criteria:

1. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.
2. Any metastasis no located in liver (liver tumor extended without discontinuity to other regional structures are accepted, see inclusion criteria).
3. Pregnancy or breast feeding (women of child-bearing potential).
4. Comorbidity with a grave prognosis (estimated survival <3 months) and/or worse then the basic disease for which the patients will be included in the study.
5. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
6. Patients who are declared incompetent.
7. Female patients who are not using an acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) OR are less than 1 year postmenopausal or surgically sterile during their participation in this study (from the time they sign the consent form) to prevent pregnancy.
8. Active hepatitis (B and/or C).
9. Allergy for I.V. contrast or anesthesic agents used.
10. Scan or MRI contra-indications: severe claustrophobia, metal shrapnel, implanted pacemaker and/or neurostimulators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
size of tumor | 12 weeks
  evaluation criteria for solid tumors RECIST

SECONDARY OUTCOMES:
Progression free survival PFS | 12 weeks
  PFS-end-point was defined as either Imaging progression or death of any cause
HPFS | 12 weeks
  Hepatic free survival

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand NASSAR, MD, PhD, Study Director — AFPREMED
Locations (1):
- Tongji University Eastern Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided